CLINICAL TRIAL: NCT05869721
Title: Effects of Yoga on Physical Functioning and Sleep Quality of Women with Breast Cancer: a Pilot Randomized Controlled Trial
Brief Title: Effects of Yoga on Women with Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Shamay Ng, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023_Yoga_Breastcancer
Record Dates: First submitted 2023-05-03; First posted 2023-05-22 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Upper Limb Functions; Sleep Quality; Upper Limb Muscle Strength; Shoulder Mobility; Heart Rate Variability; Mood; Health-related Quality of Life
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Yoga

STUDY DESIGN:
Intervention Model Description: This pilot randomized controlled trial will conduct at a university-affiliated rehabilitation laboratory staring from May 2023 in Hong Kong.
Who Masked: Outcomes Assessor
Masking Description: After the baseline assessment, all eligible participants will be allocated randomly in a 1:1 ratio to either (1) experimental group which received yoga programme over a period of eight weeks, or (2) wait-list control group. The research assistant, who is responsible for allocation, is independent from the data collection and analysis, and the intervention. The participants will be reminded not to disclose information related to group allocation to the assessors to prevent possible bias during measurement. All assessments will be performed by an assessor who is blinded to the group allocation and not involved in the delivery of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Yoga group (Experimental): Participants will receive yoga programme over a period of eight weeks
  Interventions: Other: Yoga
- Control group (No Intervention): The participants in the control group will receive usual care, and complete all assessments on the same timeline as the intervention group. They will be offered yoga programme at the completion of the final measurement.

INTERVENTIONS:
Other: Yoga — The yoga forms are designed from the modified traditional Hatha yoga style consisting of pranayama, asana, meditation with additional relaxation elements. The selected postures will engage core and upper limb muscle and which proposed to strengthen the whole body, increase flexibility of shoulder and limbs, particularly, improve upper limb mobility and functions; also, the progression of the yoga therapy is targeted to reach the variations of postures. The combined relaxation elements reinforced to achieve restoration of the body so as to improve sleep.
  Arms: Yoga group

SUMMARY:
Upper limb complications and sleep disturbances are prevalent, persistent, and serious health problems in women with breast cancer. However, these problems are underrecognized in clinical practice and thus have substantial adverse impacts on the health and quality of life of women with breast cancer. As yoga practices have been shown to improve physical and psychological health in people with cancer, such practices may also alleviate upper limb complications and sleep disturbances in women with breast cancer. However, there are few evidence-based guidelines or protocols to support the integration of yoga therapy into clinical practice for managing the health conditions of women with breast cancer. Therefore, this study aims to investigate the effects of yoga therapy on improving the upper limb functions, sleep quality, and quality of life in women with breast cancer.

DETAILED DESCRIPTION:
Breast cancer is the most commonly diagnosed cancer worldwide, accounting for 12% of all new cancer cases annually, and there were an estimated 2.3 million new cases worldwide in 2020. Contemporary breast cancer treatments have improved therapeutic outcomes. However, these treatments cause adverse effects; for example, more than half of women with breast cancer experience treatment-related comorbidities.

Over 60% of women with breast cancer have reported experiencing ipsilateral upper limb complications immediately post-treatment and these complications may become chronic or permanent disorders. Upper limb dysfunction is a long-term complication that comprises a complex range of symptoms and disorders, including lymphedema, pain, decreased joint mobility and muscle strength, sensory alterations, and neuropathies. Another prevalent and persistent problem that has been reported is sleep disturbance. According to a recent review, the prevalence of sleep disturbance ranged from 14 to 90% [pooled estimated 0.4; 95% Confidence Interval (CI) 0.29 to 0.52], and the persistence rate has been found to be more than 50%. Such side effects may lead to individual suffering and economic burdens, and can compromise the quality of life of women with breast cancer. Thus, the management of treatment-related side effects is an important part of the supportive care of women with breast cancer.

Yoga is based on ancient India philosophy, and emphasizes the integration of postures, breathing, and meditation. This mind-body practice has gained popularity over the last decades and serves as a complementary approach that is commonly used for various health conditions. This safe and trendy exercise holds attractive to female target participants. Yoga combines joint movements and breathing exercises that can help the lungs to expand, resulting in the stretching of muscles and thus increasing lymphatic circulation, which improves upper limb function. Besides, Yoga combines physical activity with mindful elements consisting of breathing and meditative practices. The practice of such mindfulness with the engagement of skeletal muscles represents a holistic approach that may decrease sleep disturbance.

Upper limb complications and sleep disturbances are prevalent, persistent, and serious health problems in women with breast cancer. However, these problems are underrecognized in clinical practice and thus have substantial adverse impacts on the health and quality of life of women with breast cancer. As yoga practices have been shown to improve physical and psychological health in people with cancer, such practices may also alleviate upper limb complications and sleep disturbances in women with breast cancer. However, there are few evidence-based guidelines or protocols to support the integration of yoga therapy into clinical practice for managing the health conditions of women with breast cancer. Therefore, this study aims to investigate the effects of yoga therapy on improving the upper limb functions, sleep quality, and quality of life in women with breast cancer. The research hypothesis of this study were (1) improvements in upper limb functions and sleep quality, could be observed in the experimental group across the assessment time points and (2) the experimental group should have better upper limb performance and sleep parameters than the control group immediately after Yoga intervention and also at the follow up.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18
* Female
* Normal cognitive function
* Diagnosed with primary breast cancer of stage I-III
* Completed cancer-related treatments (including surgery, radiotherapy, and/or chemotherapy) at least 4 weeks before enrollment except conventional medical care (e.g., hormonal therapy)

Exclusion Criteria:

* Diagnosed with distant metastasis in non-breast body part
* Diagnosed with significant diseases, such as cardiovascular, respiratory, neurological, musculoskeletal (except upper-extremity problems secondary to breast cancer), endocrine, metabolic, and psychological disorders
* Being pregnant
* Prior experiences of practicing yoga

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with breast cancer (based on self-representation of gender identity)
Enrollment: 34 (Actual)
Dates: Start 2023-05-04 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Upper limb functional status, score range 0-100%, higher score means more severe disability | T1: baseline (before the study begins).
  Will be assessed using the short form of the Chinese (Hong Kong) version of the Disabilities of Arm-Shoulder-Hand Questionnaire (quickDASH-HKPWH)
Change from baseline Upper limb functional status at 4 weeks | T2: mid-intervention (week 4)
  Will be assessed using the short form of the Chinese (Hong Kong) version of the Disabilities of Arm-Shoulder-Hand Questionnaire (quickDASH-HKPWH), score range 0-100%, higher score means more severe disability
Change from baseline Upper limb functional status at 8 weeks | T3: immediately post-intervention (week 8)
  Will be assessed using the short form of the Chinese (Hong Kong) version of the Disabilities of Arm-Shoulder-Hand Questionnaire (quickDASH-HKPWH), score range 0-100%, higher score means more severe disability
Change from baseline Upper limb functional status at 12 weeks | T4: 1 month follow up (week 12)
  Will be assessed using the short form of the Chinese (Hong Kong) version of the Disabilities of Arm-Shoulder-Hand Questionnaire (quickDASH-HKPWH), score range 0-100%, higher score means more severe disability
Sleep quality | T1: baseline (before the study begins)
  Will be assessed by the Chinese (for Hong Kong) version of the Pittsburgh Sleep Quality Index questionnaire, score range 0-21, higher score means poorer sleep
Change from baseline Sleep quality at 4 weeks | T2: mid-intervention (week 4)
  Will be assessed by the Chinese (for Hong Kong) version of the Pittsburgh Sleep Quality Index questionnaire, score range 0-21, higher score means poorer sleep
Change from baseline Sleep quality at 8 weeks | T3: immediately post intervention (week 8)
  Will be assessed by the Chinese (for Hong Kong) version of the Pittsburgh Sleep Quality Index questionnaire, score range 0-21, higher score means poorer sleep
Change from baseline Sleep quality at 12 weeks | T4: 1 month follow up (week 12)
  Will be assessed by the Chinese (for Hong Kong) version of the Pittsburgh Sleep Quality Index questionnaire, score range 0-21, higher score means poorer sleep

SECONDARY OUTCOMES:
Upper limb muscle strength | T1: baseline (before the study begins)
  Will be determined using a handheld dynamometer, measures muscle strength in kg, higher score means better muscle strength
Change from baseline Upper limb muscle strength at 4 weeks | T2: mid-intervention (week 4)
  Will be determined using a handheld dynamometer, measures muscle strength in kg, higher score means better muscle strength
Change from baseline Upper limb muscle strength at 8 weeks | T3: immediately post intervention (week 8)
  Will be determined using a handheld dynamometer, measures muscle strength in kg, higher score means better muscle strength
Change from baseline Upper limb muscle strength at 12 weeks | T4: 1 month follow up (week 12)
  Will be determined using a handheld dynamometer, measures muscle strength in kg, higher score means better muscle strength
Shoulder mobility | T1: baseline (before the study begins)
  Will be determined by measuring the active range of motion using a goniometer, measures range of movement in degree, higher score means better shoulder flexibility
Change from baseline Shoulder mobility at 4 weeks | T2: mid-intervention (week 4)
  Will be determined by measuring the active range of motion using a goniometer, measures range of movement in degree, higher score means better shoulder flexibility
Change from baseline Shoulder mobility at 8 weeks | T3: immediately post intervention (week 8)
  Will be determined by measuring the active range of motion using a goniometer, measures range of movement in degree, higher score means better shoulder flexibility
Change from baseline Shoulder mobility at 12 weeks | T4: 1 month follow up (week 12)
  Will be determined by measuring the active range of motion using a goniometer, measures range of movement in degree, higher score means better shoulder flexibility
Mood (including anxiety and depression symptoms) | T1: baseline (before the study begins)
  Will be assessed using The Cantonese/Chinese version of the Hospital Anxiety and Depression questionnaire, score range 0-21, higher score means more severe anxiety and depression
Change from baseline Mood (including anxiety and depression symptoms) at 4 weeks | T2: mid-intervention (week 4)
  Will be assessed using The Cantonese/Chinese version of the Hospital Anxiety and Depression questionnaire, score range 0-21, higher score means more severe anxiety and depression
Change from baseline Mood (including anxiety and depression symptoms) at 8 weeks | T3: immediately post intervention (week 8)
  Will be assessed using The Cantonese/Chinese version of the Hospital Anxiety and Depression questionnaire, score range 0-21, higher score means more severe anxiety and depression
Change from baseline Mood (including anxiety and depression symptoms) at 12 weeks | T4: 1 month follow up (week 12)
  Will be assessed using The Cantonese/Chinese version of the Hospital Anxiety and Depression questionnaire, score range 0-21, higher score means more severe anxiety and depression
Fatigue | T1: baseline (before the study begins)
  Will be assessed using the Chinese (Cantonese) version of the Fatigue Assessment Scale questionnaire, score range 10-50, higher score means more severe fatigue
Change from baseline Fatigue at 4 weeks | T2: mid-intervention (week 4)
  Will be assessed using the Chinese (Cantonese) version of the Fatigue Assessment Scale questionnaire, score range 10-50, higher score means more severe fatigue
Change from baseline Fatigue at 8 weeks | T3: mid-intervention (week 8)
  Will be assessed using the Chinese (Cantonese) version of the Fatigue Assessment Scale questionnaire, score range 10-50, higher score means more severe fatigue
Change from baseline Fatigue at 12 weeks | T4: 1 month follow up (week 12)
  Will be assessed using the Chinese (Cantonese) version of the Fatigue Assessment Scale questionnaire, score range 10-50, higher score means more severe fatigue
Heart rate variability | T1: baseline (before the study begins)
  Will be recorded over a 5-minute period using a validated wearable monitor
Change from baseline Heart rate variability at 4 weeks | T2: mid-intervention (week 4)
  Will be recorded over a 5-minute period using a validated wearable monitor
Change from baseline Heart rate variability at 8 weeks | T3: immediately post intervention (week 8)
  Will be recorded over a 5-minute period using a validated wearable monitor
Change from baseline Heart rate variability at 12 weeks | T4: 1 month follow up (week 12)
  Will be recorded over a 5-minute period using a validated wearable monitor
Health-related quality of Life | T1: baseline (before the study begins)
  Will be assessed by the Chinese-Traditional version of the Functional Assessment of Cancer Therapy-Lymphedema questionnaire, score range 0-148, higher score means better quality of life
Change from baseline Health-related quality of Life at 4 weeks | T2: mid-intervention (week 4)
  Will be assessed by the Chinese-Traditional version of the Functional Assessment of Cancer Therapy-Lymphedema questionnaire, score range 0-148, higher score means better quality of life
Change from baseline Health-related quality of Life at 8 weeks | T3: immediately post intervention (week 8)
  Will be assessed by the Chinese-Traditional version of the Functional Assessment of Cancer Therapy-Lymphedema questionnaire, score range 0-148, higher score means better quality of life
Change from baseline Health-related quality of Life at 12 weeks | T4: 1 month follow up (week 12)
  Will be assessed by the Chinese-Traditional version of the Functional Assessment of Cancer Therapy-Lymphedema questionnaire, score range 0-148, higher score means better quality of life

CONTACTS AND LOCATIONS:
Locations (2):
- Hong Kong (2):
  - A university-affiliated rehabilitation laboratory, Hung Hom, Kowloon
  - The Hong Kong Polytechnic University, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
The datasets of the study will only be available from the corresponding author on reasonable request after the findings being published in peer-reviewed journal.